CLINICAL TRIAL: NCT00553202
Title: Killer Immunoglobulin-like Receptor (KIR) Incompatible Unrelated Donor Hematopoietic Cell Transplantation (SCT) for AML With Monosomy 7, -5/5q-, High FLT3-ITD AR, or Refractory and Relapsed Acute Myelogenous Leukemia (AML) in Children: A Children's Oncology Group (COG) Study
Brief Title: Donor Stem Cell Transplant in Treating Young Patients With Acute Myeloid Leukemia With Monosomy 7, -5/5q-, High FLT3-ITD AR, or Refractory or Relapsed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML05P1; COG-AAML05P1 (Other: Children's Oncology Group); NCI-2009-00321 (Registry Identifier: NCI Trial Identifier)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Cyclophosphamide; Cyclosporine; Cyclosporins; Methotrexate; Methylprednisolone; Methylprednisolone Hemisuccinate; Tacrolimus; allogenic effect factor; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy and allogeneic SCT) (Experimental): Patients receive busulfan IV every 6 hours on days -9 to -6, high-dose cyclophosphamide IV over 1 hour on days -5 to -2, anti-thymocyte globulin IV once or twice daily over 4 hours on days -3 to -1, and methylprednisolone IV on days -3 to -1.
  Patients undergo allogeneic hematopoietic stem cell transplantation (SCT) or allogeneic bone marrow transplantation (BMT) on day 0.
  Patients receive cyclosporine or tacrolimus IV or orally beginning on day -2 and continuing until day 50, followed by a taper until week 24. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Blood samples will be collected periodically from both patients and donors for studies of natural killer cells in support of the pharmacological study objectives
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Drug: methylprednisolone; Drug: tacrolimus; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — Given IV
  Other Names: Rabbit ATG; RATG-Rabbit; Antithymocyte Globulin; Thymoglobulin; NSC #720095
Drug: busulfan — Given IV
  Other Names: Busulfex; NSC #750
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC #26271
Drug: cyclosporine — Given IV or orally
  Other Names: CYA; Sandimmune; Neoral; Gengraf; NSC #290193
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; NSC #000740
Drug: methylprednisolone — Given IV
  Other Names: Solu-Medrol; A-Methapred; Medrol; NSC #19987
Drug: tacrolimus — Given IV
  Other Names: FK-506; Prograf; NSC #717865
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
Procedure: allogeneic bone marrow transplantation — allogeneic bone marrow transplantation
  Other Names: bone marrow therapy; allogeneic; allogenic; transplantation; allogeneic bone marrow; allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic hematopoietic SCT

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant using stem cells that closely match the patient's stem cells, helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine, tacrolimus, and methotrexate before and after transplant may stop this from happening.

PURPOSE: Natural Killer (NK) cells from the donor's bone marrow may be important in fighting leukemia. Bone marrow donors can be selected based on the type of NK cells they have, specifically the killer immunoglobulin receptor (KIR) type. This study provides information on KIR type from potential donors, which can be used in selecting the bone marrow donor. This phase II trial of unrelated donor stem cell transplant in patients with high risk AML (monosomy 7, -5/5q-, high FLT3-ITD AR, or refractory or relapsed AML) in which KIR typing of the patients and potential donors will be available to the treating transplant physician at the time of donor selection.

DETAILED DESCRIPTION:
OBJECTIVES:

* To define the relationship between the status of donor NK-cell receptor and patient outcomes after killer immunoglobulin-like receptor-incompatible unrelated donor (URD) and umbilical cord blood (UCB) hematopoietic cell transplantation (HCT) in young patients with acute myeloid leukemia with monosomy 7, -5/5q-, high FLT3 internal tandem duplication allelic ratio (High-FLT3-ITD AR), or refractory or relapsed acute myelogenous leukemia.
* To correlate the relationships between factors affecting NK receptor status and clinical events.
* To assess NK-cell development after URD and UCB HCT in patients with poor prognosis AML.
* To evaluate NK-cell reconstitution and receptor-acquisition pattern in these patients.

OUTLINE: This is a multicenter study.

* Preparative regimen: Patients receive 1 of the following regimens:

  * Hematopoietic stem cell transplantation (SCT): Patients receive busulfan IV every 6 hours on days -9 to -6, high-dose cyclophosphamide IV over 1 hour on days -5 to -2, anti-thymocyte globulin IV once or twice daily over 4 hours on days -3 to -1, and methylprednisolone IV on days -3 to -1.
  * Umbilical cord blood (UCB) transplantation: Conditioning regimen, infusion procedures, and post-transplant immunoprophylaxis for patients with an UCB donor are according to institutional guidelines and standards.
* Allogeneic hematopoietic stem cell transplantation (SCT) or umbilical cord blood (UCB) transplant: Patients undergo allogeneic SCT or UCB transplant on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive cyclosporine or tacrolimus IV or orally beginning on day -2 and continuing until day 50, followed by a taper until week 24. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Blood samples will be collected periodically from both patients and donors for studies of natural killer cells in support of the study objectives.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Patients with primary refractory acute myeloid leukemia (AML), defined as ≥ 5% bone marrow blasts after two induction courses of chemotherapy
  * Primary refractory AML, defined as ≥ 5% bone marrow blasts after two induction courses of chemotherapy
  * AML or myelodysplastic syndrome with -5/5q- or monosomy 7 without inv(16)/t(16;16) or t(8;21) cytogenetics or NPM or CEBPα mutations
  * Relapsed AML (≥ 5% bone marrow blasts) who meet the customary WHO criteria for AML
  * AML and high FLT3 internal tandem duplication allelic ratio (high FLT3-ITD AR), defined as > 0.4
  * All cases of therapy-related AML (therapy-related AML is considered high risk)
  * Patients with AML, without inv(16)/t(16;16) or t(8;21), monosomy 7, -5/5q-, NPM, or CEPBα mutations, or high FLT3-ITD AR, but with evidence of residual AML (≥ 0.1%) at the end of Induction I; or if a minimal residual disease (MRD) is not performed, then with > 15% bone marrow blasts by morphology after one induction course of chemotherapy

    * Any flow-based MRD is eligible for AAML05P1 for patients not on AAML1031, whereas patients on AAML1031 must utilize the central lab as per the AAML1031 protocol guidelines
* No Fanconi anemia
* Recipients of unrelated marrow or cord blood are eligible for this study

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) (for patients over 16 years of age) or Lansky PS (for patients 16 and under) 50-100%
* Total bilirubin ≤ 2 mg/dL
* SGOT (AST) or SGPT (ALT) ≤ 2.5 times upper limit of normal
* DLCO ≥ 50% OR a normal chest x-ray and pulse oximetry in patients who are unable to undergo pulmonary function tests
* Shortening fraction ≥ 27% by ECHO
* Creatinine clearance or radioisotope glomerular filtration rate at least 60 mL/min OR creatinine adjusted according to age
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with proven or suspected bacterial sepsis, pneumonia, or meningitis are eligible provided appropriate therapeutic measures have been initiated to control the presumed or proven infection, and systemic signs are not life-threatening
* No evidence or presence of a fungal infection within the past 30 days

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy, radiotherapy or any antileukemic therapy allowed provided patients meet 1 of the following criteria:

  * Received initial treatment for relapsed AML
  * Patients with primary induction failure or relapse who have already received initial therapy and who may have gone on to have additional therapy prior to receiving protocol stipulated therapy on AAML05P1
* No treatment for fungal infection within the past 30 days
* Concurrent radiotherapy to localized painful lesions allowed
* No other concurrent cancer chemotherapy or immunomodulating agents

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Actual)
Dates: Start 2008-01; Primary Completion 2016-06 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stella M. Davies, MBBS, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (52):
- United States (48):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Central California, Madera, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Children's and Women's Hospital of British Columbia, Vancouver, British Columbia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy and Allogeneic SCT): All patients
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Started | 158
Completed | 90
Not Completed | 68
Not completed — Death | 16
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 28
Not completed — Withdrawal by Subject | 1
Not completed — No donor identified | 16
Not completed — Fails to meet organ function | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 149
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 3215.34 (2240.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 128
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  Canada | 11
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS - Time from HSCT until death
Time Frame: At 5 years from HSCT date
Population: Patients without completion of planned therapy (n=68) are excluded from analyses of OS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 90
Percentage of participants | 45.9 [33.7 to 57.2]

2. Primary Outcome: Cumulative Incidence of NK Cell Reconstitution
Description: Cumulative incidence of successful reconstitution to donor level is calculated.
Time Frame: At 5 years from HSCT date
Population: Patients without completion of planned therapy (n=68) or without NK cell status (n=38) are excluded from analyses of TExp
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 52
Percentage of participants | 48.1 [33.8 to 61.0]

3. Other Pre Specified Outcome: Disease-free Survival
Description: The cumulative incidence of relapse or death after SCT will be calculated by considering relapse and death due to other causes as competing events.
Time Frame: From the date of SCT to the date of relapse, the date of death, or the date of last follow-up, whichever occurs first
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Acute and Chronic Graft-versus-host Disease
Description: Acute and chronic GVHD will be summarized.
Time Frame: Up to 5 years
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Time to the Donor-specific NK-cell Receptor Expression
Description: The presence of donor cells is demonstrated by the detection of informative variable-number tandem-repeat polymorphisms or by fluorescent in situ hybridization with a Y-chromosome-specific probe in cases of sex-mismatched transplants. Independent variables that will be examined include donor-recipient KIR mismatch, taking into consideration the interactions with donor-recipient human leukocyte antigen (HLA) compatibility, and the numbers of CD34+ cells and CD3+ cells in the graft.
Time Frame: Up to 42 days after SCT
Arm/Group | Treatment (Chemotherapy and Allogeneic SCT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Group 1: All patients
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 7/90
Other Adverse Events (participants affected / at risk) | 32/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=90)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Alanine aminotransferase increased (Investigations) | 1 — Adeers submitted
Ascites (Gastrointestinal disorders) | 1 — Adeers submitted
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Blood bilirubin increased (Investigations) | 1 — Adeers submitted
Creatinine increased (Investigations) | 1 — Adeers submitted
Death NOS (General disorders) | 2 — Adeers submitted
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 — Adeers submitted
Hypercalcemia (Metabolism and nutrition disorders) | 1 — Adeers submitted
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Immune system disorders - Other, specify (Immune system disorders) | 1 — Adeers submitted
Infections and infestations - Other, specify (Infections and infestations) | 2 — Adeers submitted
Mucositis oral (Gastrointestinal disorders) | 1 — Adeers submitted
Multi-organ failure (General disorders) | 1 — Adeers submitted
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Portal hypertension (Hepatobiliary disorders) | 1 — Adeers submitted
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Adeers submitted
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 — Adeers submitted
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers submitted
Sepsis (Infections and infestations) | 2 — Adeers submitted
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=90)
Abdominal distension (Gastrointestinal disorders) | 1 — Adeers not subm
Abdominal pain (Gastrointestinal disorders) | 1 — Adeers not subm
Acute kidney injury (Renal and urinary disorders) | 5 — Adeers not subm
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers not subm
Allergic reaction (Immune system disorders) | 1 — Adeers not subm
Ascites (Gastrointestinal disorders) | 8 — Adeers not subm
Aspartate aminotransferase increased (Investigations) | 2 — Adeers not subm
Bladder spasm (Renal and urinary disorders) | 1 — Adeers not subm
Blood bilirubin increased (Investigations) | 11 — Adeers not subm
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers not subm
Cardiac disorders - Other, specify (Cardiac disorders) | 2 — Adeers not subm
Creatinine increased (Investigations) | 1 — Adeers not subm
Cystitis noninfective (Renal and urinary disorders) | 3 — Adeers not subm
Cytokine release syndrome (Immune system disorders) | 1 — Adeers not subm
Death NOS (General disorders) | 1 — Adeers not subm
Diarrhea (Gastrointestinal disorders) | 3 — Adeers not subm
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 — Adeers not subm
Encephalitis infection (Infections and infestations) | 1 — Adeers not subm
Febrile neutropenia (Blood and lymphatic system disorders) | 1 — Adeers not subm
Gastric hemorrhage (Gastrointestinal disorders) | 1 — Adeers not subm
Heart failure (Cardiac disorders) | 1 — Adeers not subm
Hematuria (Renal and urinary disorders) | 2 — Adeers not subm
Hepatic pain (Hepatobiliary disorders) | 4 — Adeers not subm
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 — Adeers not subm
Hyperglycemia (Metabolism and nutrition disorders) | 3 — Adeers not subm
Hypernatremia (Metabolism and nutrition disorders) | 2 — Adeers not subm
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 — Adeers not subm
Hypoglycemia (Metabolism and nutrition disorders) | 2 — Adeers not subm
Hypokalemia (Metabolism and nutrition disorders) | 4 — Adeers not subm
Hyponatremia (Metabolism and nutrition disorders) | 1 — Adeers not subm
Hypophosphatemia (Metabolism and nutrition disorders) | 1 — Adeers not subm
Hypotension (Vascular disorders) | 2 — Adeers not subm
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 — Adeers not subm
Ileus (Gastrointestinal disorders) | 1 — Adeers not subm
Infections and infestations - Other, specify (Infections and infestations) | 3 — Adeers not subm
Left ventricular systolic dysfunction (Cardiac disorders) | 4 — Adeers not subm
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 — Adeers not subm
Lung infection (Infections and infestations) | 1 — Adeers not subm
Mucositis oral (Gastrointestinal disorders) | 2 — Adeers not subm
Multi-organ failure (General disorders) | 2 — Adeers not subm
Pain (General disorders) | 1 — Adeers not subm
Pericardial effusion (Cardiac disorders) | 1 — Adeers not subm
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers not subm
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers not subm
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 — Adeers not subm
Portal hypertension (Hepatobiliary disorders) | 3 — Adeers not subm
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 — Adeers not subm
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 — Adeers not subm
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 — Adeers not subm
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 — Adeers not subm
Seizure (Nervous system disorders) | 1 — Adeers not subm
Sepsis (Infections and infestations) | 2 — Adeers not subm
Serum amylase increased (Investigations) | 1 — Adeers not subm
Sinus tachycardia (Cardiac disorders) | 1 — Adeers not subm
Sinusitis (Infections and infestations) | 1 — Adeers not subm
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Adeers not subm
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 — Adeers not subm
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 — Adeers not subm
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 — Adeers not subm
Urinary tract infection (Infections and infestations) | 1 — Adeers not subm
Urine output decreased (Investigations) | 2 — Adeers not subm
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 — Adeers not subm
Vascular disorders - Other, specify (Vascular disorders) | 2 — Adeers not subm
Weight gain (Investigations) | 8 — Adeers not subm
White blood cell decreased (Investigations) | 1 — Adeers not subm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.